CLINICAL TRIAL: NCT01476397
Title: ASSESSMENT OF GROWTH OF INFANTS FED FORMULA WITH PROBIOTICS
Brief Title: Probiotic Formula and Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 10.01.US.INF
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: full-term; formula-fed infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control infant formula (Active Comparator): partially hydrolyzed whey infant formula
  Interventions: Other: Control infant formula
- test infant formula (Experimental): partially hydrolyzed whey infant formula with probiotic
  Interventions: Other: Test infant formula

INTERVENTIONS:
Other: Control infant formula — partially hydrolyzed whey infant formula consumed ad libitum throughout study
  Arms: control infant formula
Other: Test infant formula — partially hydrolyzed whey formula with probiotic
  Arms: test infant formula

SUMMARY:
This is a growth study of full-term, formula-fed infants randomized to receive a partially hydrolyzed whey protein formula with and without probiotics for the first four months of life. It is hypothesized that there will be no difference in growth between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full-term
* Birth weight > 2500 and < 4500 g
* 14±3 days of age on enrollment
* Exclusively formula-fed, singleton birth
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Known or suspected cow-milk allergy
* Congenital illness or malformation that may affect infant feeding and/or growth
* Significant prenatal and/or postnatal disease
* Any readmission to hospital prior to enrollment
* Receiving prescription medication or frequent use of over the counter medications except vitamin and mineral supplements
* Has received intravenous antibiotic therapy or oral probiotic in the last 7 days
* Currently participating in another clinical study
* Cannot be expected to comply with treatment

Ages: 11 Days to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
growth | 4 months
  weight gain assessed monthly

SECONDARY OUTCOMES:
other growth | 4 months
  Length, head circumference will be measured at monthly visits
adverse events | 4 months
  all adverse events will be documented throughout the study
stool characteristics | throughout study
  stool frequency, color, consistency
spit-up | throughout study
  frequency of spit-up as reported by caregivers
vomit | throughout study
  frequency of vomitting as reported by caregivers

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - North Scottsdale Pediatric Associates, Scottsdale, Arizona
  - Pediatrics & Adolescent Medicine, Marietta, Georgia
  - Kentucky Pediatric Adult Research, Bardstown, Kentucky
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - PMG Research of Bristol, Bristol, Tennessee
  - Pediatric Healthcare of Northwest Houston, Tomball, Texas
  - Advanced Pediatrics, Vienna, Virginia